CLINICAL TRIAL: NCT03648385
Title: Effects of DHEA in Pulmonary Hypertension
Acronym: EDIPHY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01HL141268 (NIH)
Record Dates: First submitted 2018-08-10; First posted 2018-08-27 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DHEA to placebo (Other): DHEA tablet (50 mg) taken by mouth once a day for 18 weeks, followed by 4 week washout period and then 1 placebo tablet taken by mouth once a day for 18 weeks
  Interventions: Drug: DHEA tablet; Other: Placebo
- Placebo to DHEA (Other): 1 placebo tablet taken by mouth once a day for 18 weeks, followed by 4 week washout period and then 1 DHEA tablet taken by mouth once a day for 18 weeks
  Interventions: Drug: DHEA tablet; Other: Placebo

INTERVENTIONS:
Drug: DHEA tablet — DHEA tablet (50 mg) taken by mouth once a day for 18 weeks. All participants in this crossover trial will receive DHEA during Treatment Period 1 or Treatment Period 2. There is a 4 week washout between Treatment Period 1 and Treatment Period 2
  Other Names: Dehydroepiandrosterone
Other: Placebo — 1 placebo tablet taken by mouth once a day for 18 weeks. All participants in this crossover trial will receive placebo during this crossover study during Treatment Period 1 or Treatment Period 2. There is a 4 week washout between Treatment Period 1 and Treatment Period 2

SUMMARY:
The goal of this crossover trial is to determine whether the study drug dehydroepiandrosterone (DHEA) improves right ventricular longitudinal strain measured by cardiac magnetic resonance imaging at 18 weeks AND 40 weeks compared to placebo and to assess side effects and safety in pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a heterogenous clinical disease characterized foremost by an abnormal increase in pulmonary artery pressure. Pulmonary vasculopathy, characterized by pathologic remodeling and vasoconstriction of the pulmonary arterioles, results in progressive dyspnea, exercise intolerance, right ventricular (RV) failure, and death. Female sex is the strongest clinical risk factor for PAH, with a 4:1 female-to-male ratio reported from the largest registry. Despite the increased risk of PAH in women, women with PAH have better survival than men. RV function is an important cause of morbidity and mortality in PAH as well as highly prevalent heart and lung diseases, but determinants of the RV response are entirely unknown. We and others have shown that female sex is associated with better RV systolic function in both health and disease, including PAH and left heart failure. Targeted PAH therapy leads to greater improvements in RVEF (demonstrated after just several months of treatment) in women as compared to men and partially explains better outcomes in women. Demonstration that DHEA has direct RV and sex-based effects will support the hypothesis that sex hormones play an important role in disease pathogenesis and provide insight into sex hormone manipulation as a treatment strategy in PAH.

The goal of this crossover trial is to correlate sex and sex hormones (particularly DHEA) to pulmonary vascular and RV phenotype differences in men and women with PAH. The study seeks to leverage a safe and available hormone treatment to gain further insight into 1) RV effects (a novel and critical end point in PH and PAH), 2) effects on two key PAH pathways in vivo and in vitro as a means for understanding sex-based differences in PAH, and 3) efficiency planning for a future Phase II parallel trial of DHEA as a novel treatment strategy in PAH.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of PAH that is 1) idiopathic, 2) heritable or 3) associated with connective tissue disease, congenital systemic-to-pulmonary shunt, porto-pulmonary hypertension, drug or toxin use.

Documentation of the following at any time prior to study entry:

* mPAP ≥ 25 mmHg at rest, pulmonary capillary wedge pressure or left ventricular end-diastolic pressure ≤ 15 mmHg, and PVR > 3 Wood units
* Pulmonary function testing documenting forced expiratory volume in one second/forced vital capacity ratio ≥ 70% predicted and total lung capacity ≥ 70% predicted
* If TLC is mildly reduced (60%<TLC%<70%), computerized tomography (HRCT or non-HRCT) documenting no significant interstitial lung disease may be used to fulfill this requirement.
* Chest tomography documenting no more than moderate parenchymal lung disease with clinician designated WHO I PAH and meeting both TLC and FEV1/FVC criteria.
* Normal or low probability V/Q scan
* If no V/Q scan is available, a CT angiogram documenting the absence of thromboembolic disease may be used, provided the subject meets diagnostic PAH criteria

Exclusion Criteria:

* Age < 18 years old
* PAH associated with human immunodeficiency virus infection
* New background PAH therapy within 12 weeks
* Significant dose change in background PAH therapy within 12 weeks.
* Untreated severe obstructive sleep apnea diagnosed by polysomnography
* Evidence of left-sided valvular disease or systolic dysfunction on echocardiogram (≥ moderate mitral or aortic disease or LV ejection fraction ≤ 50%)
* Glomerular filtration rate <40 mls/min/1.73m2
* Child-Pugh Class C cirrhosis
* Untreated hypo- or hyper-thyroidism
* Pregnant or breastfeeding
* Active or planned use of hormone supplements, oral contraceptive pills, hormonal therapies
* History of breast, ovarian, uterine, testicular or prostate cancer
* Current use of another investigational PAH therapy
* Contraindication to MRI (e.g., metal device or fragment)
* History of significant non-adherence or circumstance which would threaten ability to comply with cross-over design and study visit schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey E Ventetuolo, MD, MS, Principal Investigator — Brown University
Locations (1):
- Rhode Island Hospital Pulmonary Hypertension Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanders R, Walsh T, Baird GL, Atalay MK, Agarwal S, Arcuri D, Klinger JR, Mullin CJ, Simmons J, Singh N, Whittenhall M, Ventetuolo CE. Effects of Dehydroepiandrosterone in Pulmonary Hypertension (EDIPHY): A Randomized, Double-Blind, Placebo-Controlled Crossover Trial. medRxiv [Preprint]. 2025 Aug 2:2025.08.01.25332627. doi: 10.1101/2025.08.01.25332627. PMID 40766123

RESULTS

PARTICIPANT FLOW:
Groups:
- DHEA to Placebo: DHEA tablet (50 mg) taken by mouth once a day for 18 weeks
  DHEA tablet: DHEA tablet (50 mg) taken by mouth once a day for 18 weeks.
  Following washout period of 4 weeks. Placebo (1 tablet once a day) for 18 weeks
- Placebo to DHEA: 1 placebo tablet taken by mouth once a day for 18 weeks
  Placebo: 1 placebo tablet taken by mouth once a day for 18 weeks
  DHEA tablet: DHEA tablet (50 mg) taken by mouth once a day for 18 weeks.
Period: Overall Study
Arm/Group | DHEA to Placebo | Placebo to DHEA
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DHEA to placebo: DHEA tablet (50 mg) taken by mouth once a day for 18 weeks
  DHEA tablet: DHEA tablet (50 mg) taken by mouth once a day for 18 weeks.
  then
  Placebo: 1 placebo tablet taken by mouth once a day for 18 weeks
- Placebo to DHEA: 1 placebo tablet taken by mouth once a day for 18 weeks
  Placebo: 1 placebo tablet taken by mouth once a day for 18 weeks
  then
  DHEA tablet: DHEA tablet (50 mg) taken by mouth once a day for 18 weeks.
- Total: Total of all reporting groups
Arm/Group | DHEA to placebo | Placebo to DHEA | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 8 | 20
  >=65 years | 2 | 4 | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [38 to 55] | 54 [46 to 68] | 48 [39 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Total: Female | 10 | 2 | 12
  Total: Male | 4 | 10 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 9 | 19
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 32 [28 to 37] | 34 [28 to 36] | 32 [27 to 36]
6MWD [Median (Inter-Quartile Range); unit: meters] | 437 [391 to 477] | 420 [230 to 451] | 430 [352 to 457]
Functional Class [Count of Participants; unit: Participants] — Functional classification drives initial choice of therapy and is a major treatment goal in PAH. WHO class is derived from the New York Heart Association classification: Class I is no limitations; Class II is slight limitations in physical activity and no symptoms at rest; Class III is symptoms with minimal activity; Class IV is symptoms at rest. Clinicians will assess functional class at each study visit.
  Participants
    II | 11 | 8 | 19
    III | 3 | 4 | 7
PAH Diagnosis [Count of Participants; unit: Participants]
  Idiopathic | 5 | 5 | 10
  Heritable | 3 | 2 | 5
  Drug and Toxin | 0 | 1 | 1
  Connective Tissue Disease | 5 | 4 | 9
  Congenital Heart Disease | 1 | 0 | 1
EmPHasis10 [Median (Inter-Quartile Range); unit: units on a scale] — The EmPHasis-10 score interpretation in pulmonary hypertension (PH) is a numerical value from 0 to 50, where a higher score indicates a poorer health status and quality of life. This score is generated from a 10-item questionnaire that assesses how PH affects a patient's life, and it serves as a tool for risk stratification and monitoring patient well-being, with improved scores correlating to better exercise capacity and survival outcomes.
  units on a scale | 25 [20 to 29] | 19 [12 to 29] | 25 [18 to 29]
Mean PAP [Median (Inter-Quartile Range); unit: mmHg] — Hemodynamics from prior right and left heart catheterizations were reviewed for inclusion. Hemodynamic criteria were met within a single catheterization procedure at any time before study enrollment.
  mmHg | 43 [39 to 52] | 50 [43 to 57] | 45 [34 to 54]
N-terminal proBNP, pg/mL [Median (Inter-Quartile Range); unit: pg/mL] | 79.9 [63.3 to 193.8] | 193.2 [104.4 to 297.5] | 127.6 [67.3 to 239.8]
Right atrial pressure, mmHg [Median (Inter-Quartile Range); unit: mmHg] — Hemodynamics from prior right and left heart catheterizations were reviewed for inclusion. Hemodynamic criteria were met within a single catheterization procedure at any time before study enrollment.
  mmHg | 7 [6 to 12] | 10 [7 to 13] | 10 [7 to 13]
PAOP, mm Hg [Median (Inter-Quartile Range); unit: mmHg] — Pulmonary artery occlusion pressure. Hemodynamics from prior right and left heart catheterizations were reviewed for inclusion. Hemodynamic criteria were met within a single catheterization procedure at any time before study enrollment.
  mmHg | 11 [8 to 11] | 13 [9 to 13] | 11 [8 to 13]
PVR, Wood units [Median (Inter-Quartile Range); unit: woods units] — Hemodynamics from prior right and left heart catheterizations were reviewed for inclusion. Hemodynamic criteria were met within a single catheterization procedure at any time before study enrollment. Pulmonary vascular resistance (PVR) in a hemodynamic measure that must be above 3 woods units to qualify subject for enrollment.
  woods units | 5 [4 to 8] | 8 [6 to 11] | 6 [5 to 9]
Cardiac Index L/min/m^2 [Median (Inter-Quartile Range); unit: L/min/m^2] — Hemodynamics from prior right and left heart catheterizations were reviewed for inclusion. Hemodynamic criteria were met within a single catheterization procedure at any time before study enrollment.
  L/min/m^2 | 2.9 [2.7 to 3.5] | 2.7 [1.8 to 2.8] | 2.8 [2 to 3.5]
Short-Form 36 PCS [Median (Inter-Quartile Range); unit: units on a scale] — The SF-36 measures health-related quality of life by assessing eight domains: physical functioning, role limitations (physical and emotional), bodily pain, general health, vitality, social functioning, and mental health. SF-36 PCS refers to the physical component. To interpret, scores above 50 indicate better-than-average health-related quality of life, and scores below 50 indicate below-average health.
  units on a scale | 38 [36 to 42] | 45 [37 to 48] | 40 [36 to 46]
Short-Form 36 MCS [Median (Inter-Quartile Range); unit: units on a scale] — The SF-36 measures health-related quality of life by assessing eight domains: physical functioning, role limitations (physical and emotional), bodily pain, general health, vitality, social functioning, and mental health. SF-36 MCS refers to mental component summary. Scores above 50 indicate better-than-average health-related quality of life, and scores below 50 indicate below-average health
  units on a scale | 48 [42 to 57] | 54 [46 to 57] | 49 [43 to 57]
RV Longitudinal Strain, % [Median (Inter-Quartile Range); unit: %] — Study MRIs were performed at a core MRI facility used for research grade imaging. Measurements were made using CVI42, Circle Cardiovascular Imaging.
  % | -18.4 [-20.4 to -17] | -18.8 [-20 to -13.5] | -18.8 [-20.3 to -13.9]
RV peak global radial strain, % [Median (Inter-Quartile Range); unit: %] — RV peak global radial strain, %. Study MRIs were performed at a core MRI facility regularly used for research grade imaging. All MRI measurements were made using commercially available cardiac MRI software (CVI42, Circle Cardiovascular Imaging).
  % | 22.4 [18.6 to 26.8] | 18.9 [16.3 to 22.3] | 20 [16.9 to 25.7]
RV circumferential strain, % [Median (Inter-Quartile Range); unit: %] — Study MRIs were performed at a core MRI facility regularly used for research grade imaging. All MRI measurements were made using commercially available cardiac MRI software (CVI42, Circle Cardiovascular Imaging).
  Strain can be either positive, which indicates lengthening, or negative, indicating shortening. Values for normal circumferential strain are negative numbers.
  % | -14.8 [-16.8 to -12.3] | -12.2 [-14.2 to -11] | -13.3 [-16.3 to -11.2]
†RV radial strain, % [Median (Inter-Quartile Range); unit: %] — Right ventricular radial strain. Study MRIs were performed at a core MRI facility on a single Siemens 1.5T Aera with full Advanced Cardiac Package and XQ Gradients (45 mT/m @ 200 T/m/s) regularly used for research grade imaging. All MRI measurements were made using commercially available cardiac MRI software (CVI42, Circle Cardiovascular Imaging). By convention strain can be either positive, which indicates lengthening, or negative, which indicates shortening. Values for normal circumferential and longitudinal strain are negative numbers, whereas those for radial strain are positive.
  % | 22.4 [18.6 to 26.8] | 18.9 [16.3 to 22.3] | 20 [16.9 to 25.7]
RVEF, % [Median (Inter-Quartile Range); unit: %] — Right ventricular ejection fraction. A normal RVEF is 40% to 50% or higher. Lower RVEF indicates right heart dysfunction. Values below 40-45% are often considered reduced, with RVEF below 20% having a particularly strong association with worse outcomes.
  Study MRIs were performed at a core MRI facility on a single Siemens 1.5T Aera with full Advanced Cardiac Package. All MRI measurements were made using commercially available cardiac MRI software (CVI42, Circle Cardiovascular Imaging). Normal Values (Female): RV EF%: 47-80%. Normal values (Male):RV EF%: 47-74%
  % | 55 [51 to 58] | 51 [44 to 57] | 53 [48 to 57]
RVEDV, mL [Median (Inter-Quartile Range); unit: mL] — RVEDV (Right Ventricular End-Diastolic Volume) represents the volume of blood in the right ventricle at the end of its filling phase (end-diastole).Study MRIs were performed at a core MRI facility regularly used for research grade imaging. All MRI measurements were made using commercially available cardiac MRI software (CVI42, Circle Cardiovascular Imaging). Normal values (female) RVEDV: 58-154 ml (48-87 ml/m2), Normal values (Male) RV EDV: 88-227 ml (55-105 ml/m2)
  mL | 147 [123 to 182] | 181 [125 to 201] | 163 [123 to 195]
RVESV, mL [Median (Inter-Quartile Range); unit: mL] — Right Ventricular End-Systolic Volume.
  Study MRIs were performed at a core MRI facility on a single Siemens 1.5T Aera with full Advanced Cardiac Package and XQ Gradients (45 mT/m @ 200 T/m/s) regularly used for research grade imaging. All MRI measurements were made using commercially available cardiac MRI software (CVI42, Circle Cardiovascular Imaging). Normal Values (Female) RV ESV: 12-68 ml (11.0-27.6 ml/m2). Normal value (Male): RV ESV: 23-103 ml (15.4-42.9 ml/m2)
  mL | 62 [53 to 85] | 92 [55 to 114] | 71 [53 to 113]
RV stroke volume, mL [Median (Inter-Quartile Range); unit: mL] — Right ventricular stroke volume. Study MRIs were performed at a core MRI facility on a single Siemens 1.5T Aera with full Advanced Cardiac Package and XQ Gradients (45 mT/m @ 200 T/m/s) regularly used for research grade imaging. All MRI measurements were made using commercially available cardiac MRI software (CVI42, Circle Cardiovascular Imaging).
  mL | 82 [70 to 95] | 83 [69 to 97] | 82 [68 to 95]
RV mass, g [Median (Inter-Quartile Range); unit: grams] — Right ventricular mass. Study MRIs were performed at a core MRI facility on a single Siemens 1.5T Aera with full Advanced Cardiac Package and XQ Gradients (45 mT/m @ 200 T/m/s) regularly used for research grade imaging. All MRI measurements were made using commercially available cardiac MRI software (CVI42, Circle Cardiovascular Imaging).
  grams | 55 [39 to 88] | 55 [40 to 78] | 55 [39 to 88]

OUTCOME MEASURES:

1. Primary Outcome: Change in Right Ventricular (RV) Longitudinal Strain, % Cardiac Magnetic Resonance Imaging (MRI)
Description: Longitudinal strain is determined using standard cine imaging and Tissue Tracking (Strain) software (Tissue Tracking plugin, Circle Cardiovascular Imaging). Study MRIs were performed at a core MRI facility on a single Siemens 1.5T Aera with full Advanced Cardiac Package and XQ Gradients (45 mT/m @ 200 T/m/s) used for research grade imaging. 2D RV longitudinal strain: Measured from RV free wall of 4-chamber view cine CMR image. RV wall is divided into 6 equal segments. Strain can be either positive, which indicates lengthening, or negative, which indicates shortening. Normal circumferential and longitudinal strain are negative numbers, those for radial strain are positive.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Population: All patients receive both DHEA and placebo during this crossover study. One group received DHEA first, followed by a washout period, then placebo. The second group received placebo first, followed by a washout period, then DHEA.
Measure: Median (95% Confidence Interval); unit: % Change in RV Longitudinal Strain
Groups:
- DHEA to Placebo, Baseline: DHEA to Placebo group, Baseline
- Placebo to DHEA, Baseline: Placebo to DHEA group, Baseline
- DHEA to placebo, 18 Weeks: Treatment period 1: DHEA to Placebo group, measurement of % change at 18 Weeks
- Placebo to DHEA, 18 Weeks: Treatment period 1: Placebo to DHEA group, % change at 18 Weeks
- DHEA to Placebo, 40 Weeks: Treatment period 2: DHEA to Placebo group, % change between 18 and 40 Weeks
- Placebo to DHEA, 40 weeks: Treatment period 2: Placebo to DHEA group, % change between 18 and 40 Weeks
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to placebo, 18 Weeks | Placebo to DHEA, 18 Weeks | DHEA to Placebo, 40 Weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
% Change in RV Longitudinal Strain | -16.8 [-21.36 to -12.18] | -16.9 [-19.06 to -14.68] | -17.7 [-19.9 to -15.5] | -18.3 [-20.5 to -16] | -17.2 [-19.7 to -14.7] | -16.7 [-19.1 to -14.3]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks; Treatment period 1: DHEA to Placebo group, measurement of % change at 18 Weeks Treatment period 1: Placebo to DHEA group, % change at 18 Weeks; Test type: Superiority; p = 0.83, generalized estimating equations (GEE) w
Statistical Analysis 2: Comparison: DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks vs DHEA to Placebo, 40 Weeks vs Placebo to DHEA, 40 weeks; Treatment period 2: DHEA to Placebo group, % change between 18 and 40 Weeks Treatment period 2: Placebo to DHEA group, % change between 18 and 40 Weeks; Test type: Superiority; p = 0.56, generalized estimating equations (GEE) w

2. Primary Outcome: Change in Right Ventricular (RV) †RV Radial Strain, %,
Description: †Short axis, RV radial strain, % by Cardiac Magnetic Resonance Imaging (MRI). Study MRIs were performed at a core MRI facility on a single Siemens 1.5T Aera with full Advanced Cardiac Package and XQ Gradients (45 mT/m @ 200 T/m/s) used for research grade imaging. Measurements were made using CVI42, Circle Cardiovascular Imaging. 2D RV longitudinal strain: Measured from RV free wall of 4-chamber view cine CMR image. RV wall is divided into 6 equal segments. Strain can be either positive, which indicates lengthening, or negative, which indicates shortening. Normal circumferential and longitudinal strain are negative numbers, those for radial strain are positive.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: % Change in RV radial strain
Groups:
- DHEA to Placebo Baseline: DHEA to Placebo group, Baseline
Arm/Group | DHEA to Placebo Baseline | Placebo to DHEA, Baseline | DHEA to placebo, 18 Weeks | Placebo to DHEA, 18 Weeks | DHEA to Placebo, 40 Weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
% Change in RV radial strain | 22.2 [18.7 to 25.66] | 19.1 [16.03 to 22.06] | 21.1 [18.1 to 24] | 20.7 [16.7 to 24.6] | 19.3 [16.5 to 22.2] | 23.1 [19.5 to 26.7]
Statistical Analysis 1: Comparison: DHEA to Placebo Baseline vs Placebo to DHEA, Baseline vs DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.08, generalized estimating equations (GEE) w
Statistical Analysis 2: Comparison: DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks vs DHEA to Placebo, 40 Weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.03, generalized estimating equations (GEE); with sandwich estimation to correct for model misspecification

3. Primary Outcome: †RV Circumferential Strain, %
Description: Circumferential strain is determined using standard cine imaging and Tissue Tracking (Strain) software (Tissue Tracking plugin, Circle Cardiovascular Imaging). Cardiac Study MRIs were performed at a core MRI facility on a single Siemens 1.5T Aera with full Advanced Cardiac Package and XQ Gradients (45 mT/m @ 200 T/m/s) used for research grade imaging. Measurements were made using CVI42, Circle Cardiovascular Imaging. 2D RV circumferential strain: Measured from RV free wall of 4-chamber view cine CMR image. RV wall is divided into 6 equal segments. Strain can be either positive, which indicates lengthening, or negative, which indicates shortening. Normal circumferential and longitudinal strain are negative numbers, those for radial strain are positive.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: % Change in RV circumferential strain
Arm/Group | DHEA to placebo, Baseline | Placebo to DHEA, Baseline | DHEA to placebo, 18 Weeks | Placebo to DHEA, 18 Weeks | DHEA to Placebo, 40 Weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
% Change in RV circumferential strain | -14.3 [-15.94 to -12.58] | -12.3 [-13.93 to -10.63] | -13.7 [-15.2 to -12.2] | -13.3 [-15.5 to -12.2] | -12.8 [-14.4 to -11.3] | -14.4 [-16.2 to -12.6]
Statistical Analysis 1: Comparison: DHEA to placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.047, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks vs DHEA to Placebo, 40 Weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.052, generalized estimating equations (GEE)

4. Primary Outcome: RV End Diastolic Volume (RVEDV), mL
Description: % Change in RV End Diastolic Volume (RVEDV), mL by Cardiac Magnetic Resonance Imaging (MRI), strain from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups: DHEA to Placebo (DHEA taken first, followed by washout and then Placebo) and Placebo to DHEA (placebo taken first, followed by washout and then DHEA). Short-axis steady state free precession (SSFP) imaging was obtained from the base of the heart through the apex. The endocardial and epicardial borders of both ventricles are be traced manually on short axis cine images at end-diastole and end-systole with exclusion of the papillary muscles and trabeculae. EDV and ESV are calculated using Simpson's rule by summation of areas on each slice multiplied by the sum of slice thickness and image gap.
Time Frame: 18 Weeks, 40 Weeks
Measure: Median (95% Confidence Interval); unit: mL
Groups:
- DHEA to Placebo, Baseline: DHEA to Placebo group, Baseline measurement
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
mL | 156.7 [133.70 to 183.86] | 173.8 [140.19 to 215.47] | 160.4 [137.3 to 187.4] | 159.8 [130.1 to 196.3] | 161.4 [134.9 to 193.1] | 161.3 [129.8 to 200.4]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.044, generalized estimating equations (GEE) w
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.96, generalized estimating equations (GEE)

5. Primary Outcome: Change in RV Ejection Fraction Measured by Cardiac MRI
Description: Change in RV ejection fraction measured by Cardiac Magnetic Resonance Imaging (MRI), % Change in strain from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups: DHEA to Placebo (DHEA taken first, followed by washout and then Placebo) and Placebo to DHEA (placebo taken first, followed by washout and then DHEA). Short-axis steady state free precession (SSFP) imaging from the base of the heart through the apex. Ventricular EFs are calculated by dividing respective stroke volumes (EDV-ESV) by EDVs.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: % Change in RV ejection fraction
Groups:
- Placebo to DHEA, Baseline: Placebo to DHEA group, Baseline measurement
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
% Change in RV ejection fraction | 52.1 [47 to 57.1] | 49.4 [43.9 to 55.0] | 52.6 [47.0 to 58.2] | 50.3 [44.8 to 55.7] | 50.7 [46.1 to 55.4] | 49.2 [43.8 to 54.6]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.91, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.61, generalized estimating equations (GEE) w

6. Primary Outcome: RVESV, mL
Description: Change in right ventricular end-systolic volume from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups: DHEA to Placebo (DHEA taken first, followed by washout and then Placebo) and Placebo to DHEA (placebo taken first, followed by washout and then DHEA). Short-axis steady state free precession (SSFP) imaging was obtained from the base of the heart through the apex. The endocardial and epicardial borders of both ventricles are be traced manually on short axis cine images at end-diastole and end-systole with exclusion of the papillary muscles and trabeculae. EDV and ESV are calculated using Simpson's rule by summation of areas on each slice multiplied by the sum of slice thickness and image gap.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: mL
Groups:
- DHEA to Placebo group, Baseline: DHEA to Placebo group, Baseline measurement
Arm/Group | DHEA to Placebo group, Baseline | Placebo to DHEA, Baseline | DHEA to placebo, 18 Weeks | Placebo to DHEA, 18 Weeks | DHEA to Placebo, 40 Weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
mL | 73.6 [57.4 to 94.4] | 86.6 [65.6 to 114.26] | 74.2 [57.6 to 95.7] | 78.1 [59.3 to 102.9] | 78.2 [60.7 to 100.9] | 81.1 [61.7 to 106.6]
Statistical Analysis 1: Comparison: DHEA to Placebo group, Baseline vs Placebo to DHEA, Baseline vs DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.14, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks vs DHEA to Placebo, 40 Weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.84, generalized estimating equations

7. Primary Outcome: RV Stroke Volume, mL
Description: Change in Right ventricular stroke volume by cardiac MRI from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups: DHEA to Placebo (DHEA taken first, followed by washout and then Placebo) and Placebo to DHEA (placebo taken first, followed by washout and then DHEA). Stroke volume is calculated through breath-hold through-plane phase contrast imaging with a velocity encoding gradient (VENC) of <120 cm/s (larger if aliasing present) in the main PA ~2-3 cm above the pulmonary valve plane, with imaging plane oriented orthogonal to the main PA. Free-breathing phase contrast imaging in the same plane and VENC with averaging over 4 respiratory cycles.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
mL | 80.1 [73.7 to 87] | 83.9 [68.64 to 102.60] | 81.6 [72 to 92.3] | 80.3 [66.9 to 96.3] | 80.9 [70.9 to 92.4] | 77.7 [62.9 to 95.9]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.36, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.71, generalized estimating equations

8. Primary Outcome: RV Mass, g
Description: Right ventricular mass, Change in RV mass from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups: DHEA to Placebo (DHEA taken first, followed by washout and then Placebo) and Placebo to DHEA (placebo taken first, followed by washout and then DHEA). Short-axis steady state free precession (SSFP) imaging from the base of the heart through the apex. RV mass is determined at the end-diastole phase as the difference between end-diastolic epicardial and endocardial volumes X heart specific gravity (1.05 g/cm3).
Time Frame: 18 weeks, 40 weeks
Measure: Median (95% Confidence Interval); unit: g
Groups:
- DHEA to Placebo Baseline: DHEA to Placebo group, Baseline measurement
- Placebo to DHEA Baseline: Placebo to DHEA group, Baseline measurement
Arm/Group | DHEA to Placebo Baseline | Placebo to DHEA Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
g | 58.8 [46.16 to 74.9] | 55.7 [44.66 to 69.4] | 58.2 [45.2 to 74.9] | 52.2 [42.3 to 64.4] | 55.9 [45.1 to 69.3] | 54.1 [42.4 to 69.2]
Statistical Analysis 1: Comparison: DHEA to Placebo Baseline vs Placebo to DHEA Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.55, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.44, generalized estimating equations

9. Secondary Outcome: Change in Six Minute Walk Distance (6MWD) Between DHEA and Placebo
Description: Change in 6MWD from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: meters
Groups:
- DHEA to Placebo, Baseline: DHEA to Placebo, Baseline measurement
- DHEA to placebo, 18 Weeks: Treatment period 1: DHEA to Placebo group, change at 18 Weeks
- Placebo to DHEA, 18 Weeks: Treatment period 1: Placebo to DHEA group, change at 18 Weeks
- DHEA to Placebo, 40 Weeks: Treatment period 2: DHEA to Placebo group, change between 18 and 40 Weeks
- Placebo to DHEA, 40 weeks: Treatment period 2: Placebo to DHEA group, change between 18 and 40 Weeks
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to placebo, 18 Weeks | Placebo to DHEA, 18 Weeks | DHEA to Placebo, 40 Weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
meters | 433.58 [375.4 to 500.7] | 355.2 [266.8 to 472.9] | 428.3 [379.2 to 483.9] | 356.2 [263.4 to 481.7] | 402.1 [323.0 to 500.4] | 364.6 [268.6 to 495.0]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks; Treatment period 1: DHEA to Placebo group, change at 18 Weeks Treatment period 1: Placebo to DHEA group, change at 18 Weeks; Test type: Superiority; p = 0.79, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks vs DHEA to Placebo, 40 Weeks vs Placebo to DHEA, 40 weeks; Treatment period 2: DHEA to Placebo group, change between 18 and 40 Weeks Treatment period 2: Placebo to DHEA group, change between 18 and 40 Weeks; Test type: Superiority; p = 0.34, generalized estimating equations (GEE)

10. Secondary Outcome: Change in World Health Organization (WHO) Functional Class
Description: Change in WHO Functional Class (I - IV with IV indicating worse symptoms) between DHEA and placebo.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | DHEA to Placebo Baseline | Placebo to DHEA Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
score on a scale | 2.2 [2.0 to 2.4] | 2.3 [2.1 to 2.6] | 2.2 [2.0 to 2.4] | 2.4 [2.1 to 2.7] | 2.1 [1.8 to 2.4] | 2.3 [2.1 to 2.6]
Statistical Analysis 1: Comparison: DHEA to Placebo Baseline vs Placebo to DHEA Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.33, generalized estimating equations (GEE) w
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.99, generalized estimating equations (GEE) w

11. Secondary Outcome: Change in Short Form-36 Summary Scores for Physical and Mental Components
Description: Change in Short Form-36 summary scores for physical and mental components (range 0 - 100, higher scores indicating better quality of life).
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: score on a scale
Groups:
- DHEA to Placebo Baseline; DHEA to Placebo, 18 Weeks; DHEA to Placebo, 40 weeks: DHEA tablet (50 mg) taken by mouth once a day for 18 weeks
  DHEA tablet: DHEA tablet (50 mg) taken by mouth once a day for 18 week
  then
  Placebo: 1 placebo tablet taken by mouth once a day for 18 weeks
- Placebo to DHEA Baseline; Placebo to DHEA, 18 weeks; Placebo to DHEA, 40 weeks: 1 placebo tablet taken by mouth once a day for 18 weeks
  Placebo: 1 placebo tablet taken by mouth once a day for 18 weeks
  then
  DHEA tablet: DHEA tablet (50 mg) taken by mouth once a day for 18 week
Arm/Group | DHEA to Placebo Baseline | Placebo to DHEA Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
score on a scale
  SF-36, PCS | 39.4 [36.0 to 42.7] | 42.8 [38.4 to 47.2] | 39.7 [36.2 to 43.1] | 38.9 [32.6 to 45.3] | 37.0 [32.2 to 41.8] | 41.7 [37.0 to 46.4]
  SF-36, MCS | 45.1 [37.1 to 53.1] | 49.1 [41.8 to 56.3] | 43.6 [37.1 to 50.2] | 46.2 [39.5 to 53.0] | 45.2 [38.8 to 51.5] | 47.9 [40.8 to 54.9]
Statistical Analysis 1: Comparison: DHEA to Placebo Baseline vs Placebo to DHEA Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; SF-36 PCS; Test type: Superiority — Treatment period 1: DHEA to Placebo group, change at 18 Weeks Treatment period 1: Placebo to DHEA group, change at 18 Weeks; p = 0.13, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; SF-36 PCS; Test type: Superiority — Treatment period 2: DHEA to Placebo group, change between 18 and 40 Weeks Treatment period 2: Placebo to DHEA group, change between 18 and 40 Weeks; p = 0.044, generalized estimating equations (GEE)
Statistical Analysis 3: Comparison: DHEA to Placebo Baseline vs Placebo to DHEA Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; SF-36 MCS; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.77, generalized estimating equations (GEE)
Statistical Analysis 4: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; SF-MCS; Test type: Superiority — [test comment as in outcome 11, analysis 2]; p = 0.98, generalized estimating equations (GEE)

12. Secondary Outcome: Change in emPHasis-10
Description: Change in emPHasis-10 score (range 0 - 50, higher scores indicating worse quality of life) between DHEA and placebo.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | DHEA to Placebo Baseline | Placebo to DHEA Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
score on a scale | 25.4 [20.8 to 29.9] | 21.7 [13.9 to 29.5] | 25.5 [20.7 to 30.3] | 22.7 [16.1 to 29.4] | 27.3 [21.0 to 33.6] | 18.1 [11.8 to 24.3]
Statistical Analysis 1: Comparison: DHEA to Placebo Baseline vs Placebo to DHEA Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.70, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.037, generalized estimating equations (GEE)

13. Secondary Outcome: Change in NT-proBNP Between DHEA and Placebo
Description: Change in serum level of NT-proBNP between DHEA and placebo.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to placebo, 18 Weeks | Placebo to DHEA, 18 Weeks | DHEA to Placebo, 40 Weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
pg/mL | 106.8 [75.5 to 151.2] | 205.9 [105.8 to 400.6] | 156.4 [103.5 to 236.2] | 139.3 [70.0 to 289.9] | 170.3 [88.5 to 327.7] | 146.9 [77.2 to 279.9]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.005, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to placebo, 18 Weeks vs Placebo to DHEA, 18 Weeks vs DHEA to Placebo, 40 Weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.9, generalized estimating equations (GEE)

14. Secondary Outcome: Change in DHEA-S (ug/dL)
Description: Change in DHEA-S from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: ug/dL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
ug/dL | 77.8 [49.0 to 123.8] | 48.2 [26.6 to 87.5] | 287.8 [197.5 to 419.3] | 49.3 [28.2 to 86.1] | 75.9 [55.0 to 104.6] | 169.9 [87.0 to 332.0]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.034, generalized estimating equations (GEE)

15. Secondary Outcome: Change in Estradiol, pg/mL
Description: Change in Estradiol, pg/mL from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
pg/mL | 46.3 [22.9 to 93.6] | 26.3 [13.9 to 49.7] | 60.7 [33 to 111.7] | 24.7 [11.2 to 54.3] | 34.5 [18 to 66.3] | 25.3 [14.3 to 44.8]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; Treatment period 1: DHEA to Placebo group, change at 18 Weeks Treatment period 1: Placebo to DHEA group, at 18 Weeks; Test type: Superiority; p = 0.36, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.23, generalized estimating equations (GEE)

16. Secondary Outcome: Change in Testosterone, ng/dL
Description: Change in Testosterone, ng/dL from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: ng/dL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
ng/dL | 23.8 [9 to 62.7] | 10.2 [3.8 to 27.3] | 65.6 [37.3 to 115.4] | 10.4 [3.7 to 29.3] | 27 [10.8 to 67.4] | 35.3 [14.2 to 87.7]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.002, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p < 0.0001, generalized estimating equations (GEE)

17. Secondary Outcome: Change in Progesterone, ng/mL
Description: Change in Progesterone, ng/mL from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: ng/mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
ng/mL | 0.6 [0.4 to 1] | 0.6 [0.3 to 1.3] | 0.6 [0.3 to 0.9] | 0.4 [0.3 to 0.6] | 0.8 [0.4 to 1.6] | 0.4 [0.2 to 0.6]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.42, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.28, generalized estimating equations (GEE)

18. Secondary Outcome: Change in Follicle Stimulating Hormone (FSH), mIU/mL
Description: Change in FSH, mIU/mL from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: mIU/mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
mIU/mL | 11.3 [6.7 to 18.9] | 21.5 [11.8 to 39.1] | 9.7 [5.7 to 16.6] | 23.5 [13 to 42.7] | 9.4 [5.4 to 16.7] | 25.5 [14.7 to 44.2]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.08, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.65, generalized estimating equations (GEE)

19. Secondary Outcome: Change in Sex Hormone Binding Globulin (SHBG), Nmol/L
Description: Change in SHBG, nmol/L from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: nmol/L
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
nmol/L | 57.8 [41.7 to 79.9] | 61 [44.2 to 84.21] | 50.2 [38.1 to 66.1] | 62.2 [44.2 to 87.4] | 59.3 [43.1 to 81.6] | 48 [34.2 to 67.5]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.07, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p < 0.01, generalized estimating equations (GEE)

20. Secondary Outcome: Change in Luteinizing Hormone, mIU/mL
Description: Change in Luteinizing hormone, mIU/mL from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: mIU/mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
mIU/mL | 12.5 [7.9 to 12.5] | 14.3 [8.4 to 24.3] | 10.3 [6.3 to 16.7] | 14.5 [8.3 to 25.4] | 8.6 [4.7 to 15.6] | 17.5 [11.8 to 26.1]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; Treatment period 1: DHEA to Placebo group, measurement of change at 18 Weeks Treatment period 1: Placebo to DHEA group, change at 18 Weeks; Test type: Superiority; p = 0.27, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.26, generalized estimating equations (GEE)

21. Secondary Outcome: Change in Prolactin, μIU/mL
Description: Change in Prolactin, μIU/mL from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: μIU/mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
μIU/mL | 329.5 [274.8 to 395.1] | 287.8 [206.4 to 401.1] | 327.4 [256.2 to 418.2] | 293.8 [212.6 to 406.1] | 305.2 [267.3 to 348.5] | 271.4 [190.1 to 387.6]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.81, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.94, generalized estimating equations (GEE)

22. Secondary Outcome: Change in C-peptide, ng/mL
Description: Change in C-peptide, ng/mL from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: ng/mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
ng/mL | 3.3 [2.5 to 4.5] | 3.6 [2.5 to 5.3] | 3.1 [2.3 to 4.1] | 3.3 [2.3 to 4.7] | 3 [2.3 to 4.0] | 3.4 [2.5 to 4.6]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.93, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.83, generalized estimating equations (GEE)

23. Secondary Outcome: Change in Insulin, μU/mL
Description: Change in Insulin, μU/mL from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: μU/mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
μU/mL | 11.4 [7.5 to 17.4] | 13.2 [7.5 to 23.4] | 10.7 [6.7 to 17] | 12.1 [7.2 to 20.2] | 10.8 [7.1 to 16.4] | 13.5 [8 to 22.8]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.85, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.74, generalized estimating equations (GEE)

24. Secondary Outcome: Cortisol, μg/dL^2
Description: Change in Cortisol, μg/dL^2 (micrograms per deciliter squared) from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (95% Confidence Interval); unit: μg/dL^2
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
μg/dL^2 | 11.7 [8.9 to 15.4] | 9.1 [6.8 to 12.1] | 9.2 [6.7 to 12.8] | 12.6 [10.3 to 15.4] | 12.9 [9.9 to 16.6] | 11.7 [9.7 to 14.4]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.004, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; Test type: Superiority; p = 0.05, generalized estimating equations (GEE)

25. Secondary Outcome: Left Ventricular Ejection Fraction, %
Description: Change in left ventricular ejection fraction (%) measured by Cardiac Magnetic Resonance Imaging (MRI). Change in LVEG from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups: DHEA to Placebo (DHEA taken first, followed by washout and then Placebo) and Placebo to DHEA (placebo taken first, followed by washout and then DHEA). Short-axis steady state free precession (SSFP) imaging from the base of the heart through the apex was used.. Ventricular EFs are calculated by dividing respective stroke volumes (EDV-ESV) by EDVs. Normal Values: 56-78% for both males and females.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (Inter-Quartile Range); unit: % Change in LVEF
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
% Change in LVEF | 66.2 [58.3 to 73.3] | 71.8 [67.2 to 75.9] | 69.1 [65.4 to 72.6] | 71.4 [66.5 to 75.8] | 68.4 [65 to 71.7] | 73.4 [68.6 to 77.6]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.33, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.23, generalized estimating equations

26. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV) (mL)
Description: Change in left ventricular LVEDV measured by Cardiac Magnetic Resonance Imaging (MRI). Change in LVEDV from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups: DHEA to Placebo (DHEA taken first, followed by washout and then Placebo) and Placebo to DHEA (placebo taken first, followed by washout and then DHEA). Short-axis steady state free precession (SSFP) imaging was obtained from the base of the heart through the apex. The endocardial and epicardial borders of both ventricles are be traced manually on short axis cine images at end-diastole and end-systole with exclusion of the papillary muscles and trabeculae. EDV and ESV are calculated using Simpson's rule by summation of areas on each slice multiplied by the sum of slice thickness and image gap. Normal values (Male):77-195 ml. Normal values (female):58-154 ml.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
mL | 104.9 [94.8 to 116.1] | 109.9 [95.5 to 126.4] | 107.7 [94.8 to 122.4] | 102.7 [87 to 121.3] | 105.3 [90.7 to 122.3] | 101 [87.2 to 117.1]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.19, generalized estimating equations (GEE)
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.94, generalized estimating equations (GEE)

27. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV) (mL)
Description: Change in LVESV measured by Cardiac Magnetic Resonance Imaging (MRI). Change in LVEDV from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups: DHEA to Placebo (DHEA taken first, followed by washout and then Placebo) and Placebo to DHEA (placebo taken first, followed by washout and then DHEA). Short-axis steady state free precession (SSFP) imaging was obtained from the base of the heart through the apex. The endocardial and epicardial borders of both ventricles are be traced manually on short axis cine images at end-diastole and end-systole with exclusion of the papillary muscles and trabeculae. EDV and ESV are calculated using Simpson's rule by summation of areas on each slice multiplied by the sum of slice thickness and image gap. Normal Values (Female):13-51 ml. Normal values (Male):19-72 ml
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
mL | 31 [25.8 to 37.2] | 31.4 [23.7 to 41.5] | 32.7 [26.7 to 40] | 30.5 [22.1 to 42.1] | 32.5 [25.8 to 41.1] | 26.1 [19.9 to 34.4]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.62, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.39, generalized estimating equations (GEE)

28. Secondary Outcome: Left Ventricular Stroke Volume (mL)
Description: Change in Left ventricular stroke volume measured by Cardiac Magnetic Resonance Imaging (MRI). Change in Left ventricular stroke volume from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups: DHEA to Placebo (DHEA taken first, followed by washout and then Placebo) and Placebo to DHEA (placebo taken first, followed by washout and then DHEA).
  Stroke volume is calculated through breath-hold through-plane phase contrast imaging with a velocity encoding gradient (VENC) of <120 cm/s (larger if aliasing present) in the main PA ~2-3 cm above the pulmonary valve plane, with imaging plane oriented orthogonal to the main PA. Free-breathing phase contrast imaging in the same plane and VENC with averaging over 4 respiratory cycles.
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
mL | 72.8 [66.8 to 79.3] | 78.4 [68.0 to 90.4] | 74.0 [65.9 to 83.2] | 75.5 [65.7 to 86.6] | 71.5 [62.6 to 81.6] | 72.2 [62.6 to 83.2]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.33, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.88, generalized estimating equations (GEE)

29. Secondary Outcome: Left Ventricular End Diastolic Mass, g
Description: Change in Left ventricular end diastolic mass, g measured by Cardiac Magnetic Resonance Imaging (MRI). Change in Left ventricular end diastolic mass, g from baseline to 18 weeks (treatment period 1) and 18 week to 40 weeks (treatment period 2) in both groups: DHEA to Placebo (DHEA taken first, followed by washout and then Placebo) and Placebo to DHEA (placebo taken first, followed by washout and then DHEA). Short-axis steady state free precession (SSFP) imaging from the base of the heart through the apex. LV mass is determined at the end-diastole phase as the difference between end-diastolic epicardial and endocardial volumes X heart specific gravity (1.05 g/cm3).
Time Frame: Baseline to 18 weeks (treatment period 1), 18 weeks to 40 weeks (treatment period 2)
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | DHEA to Placebo, Baseline | Placebo to DHEA, Baseline | DHEA to Placebo, 18 Weeks | Placebo to DHEA, 18 weeks | DHEA to Placebo, 40 weeks | Placebo to DHEA, 40 weeks
Number analyzed (Participants) | 14 | 12 | 14 | 12 | 14 | 12
g | 117.8 [97 to 143] | 119.3 [102.5 to 138.9] | 122.2 [104.3 to 143.2] | 119.5 [104.5 to 136.6] | 116.6 [98.8 to 137.7] | 114 [100.2 to 129.7]
Statistical Analysis 1: Comparison: DHEA to Placebo, Baseline vs Placebo to DHEA, Baseline vs DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.55, generalized estimating equations
Statistical Analysis 2: Comparison: DHEA to Placebo, 18 Weeks vs Placebo to DHEA, 18 weeks vs DHEA to Placebo, 40 weeks vs Placebo to DHEA, 40 weeks; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 1.00, generalized estimating equations (GEE)

30. Secondary Outcome: Treatment-related Side Effects and Adverse Events
Description: Treatment-related side effects and adverse events (as assessed by CTCAE v4.0). All participants in this trial received both DHEA and Placebo during the trial, therefore, side-effects and adverse events are listed according to the treatment or washout period in which they occurred.
Time Frame: 18 weeks, 40 weeks
Population: Data shown as n (%) of all adverse events during DHEA, placebo or the washout period. Includes only events that occurred ≥ 2 times during the study. *Specifically queried at each study visit.
Measure: Number; unit: participants
Groups:
- DHEA: Treatment group
- Placebo: Placebo Group
- Washout: Washout period
Arm/Group | DHEA | Placebo | Washout
Number analyzed (Participants) | 26 | 26 | 26
participants
  Acne | 6 | 0 | 0
  Catheter related infection | 2 | 2 | 0
  Seborrhoea | 3 | 1 | 1
  Hair Growth | 2 | 0 | 1
  Hair Loss | 0 | 2 | 0
  Headache | 1 | 0 | 1
  Diarrhea | 0 | 2 | 0
  Dizziness | 0 | 2 | 0
  Dry skin | 1 | 1 | 0
  Hypokalemia | 2 | 0 | 0
  Peripheral swelling | 0 | 1 | 1
  Pruritis | 1 | 0 | 1
  Rash | 0 | 2 | 0
  Sepsis | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at 2 weeks, 18 weeks, 19 weeks, 22 weeks, 24 weeks, 40 weeks and 42 weeks
Groups:
- DHEA: DHEA tablet (50 mg) taken by mouth once a day for 18 weeks
  DHEA tablet: DHEA tablet (50 mg) taken by mouth once a day for 18 weeks.
- Placebo: 1 placebo tablet taken by mouth once a day for 18 weeks
  Placebo: 1 placebo tablet taken by mouth once a day for 18 weeks
- DHEA Washout: Washout Period between Placebo and DHEA
- Placebo Washout: Washout Period DHEA and Placebo
Arm/Group | DHEA | Placebo | DHEA Washout | Placebo Washout
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/26 | 10/26 | 1/26 | 2/26
Other Adverse Events (participants affected / at risk) | 16/26 | 16/26 | 2/26 | 6/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DHEA (N=26) | Placebo (N=26) | DHEA Washout (N=26) | Placebo Washout (N=26)
10016450 (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 — Femoral neck fracture
10053206 (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 — Fracture displacement
10073974 (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 — Device dislocation
10056871 (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — Device Failure
10060842 (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Hypercapnic Respiratory failure
10040047 (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 — Sepsis
10020850 (Endocrine disorders) | 0 | 3 | 0 | 0 — Hyperthyroidism
10002272 (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — Anaemia
10007810 (Product Issues) | 0 | 1 | 0 | 0 — Device related infection
10038695 (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Respiratory failure
10000081 (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — Abdominal pain
10084268 (Infections and infestations) | 0 | 0 | 1 | 0 — COVID-19
10042772 (General disorders) | 1 | 0 | 0 | 0 — syncope
10002034 (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — Hospitalization due to anemia
10039911 (Nervous system disorders) | 1 | 0 | 0 | 0 — Hospitalization due to seizure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DHEA (N=26) | Placebo (N=26) | DHEA Washout (N=26) | Placebo Washout (N=26)
10000147 (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — Hair growth on chin
10000496 (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0 — Acne
10001760 (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 — Alopecia
10002856 (Psychiatric disorders) | 0 | 2 | 0 | 0 — Anxiety Attack
10003664 (Cardiac disorders) | 0 | 1 | 0 | 0 — Atrial septal defect
10003875 (Immune system disorders) | 0 | 1 | 0 | 0 — Axillary Lymph node
10003988 (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 — Back pain
10006373 (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — Onychoclasis
10007810 (Infections and infestations) | 2 | 1 | 0 | 1 — Device related infection
10007909 (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — Cellulitis
10009851 (Infections and infestations) | 1 | 2 | 0 | 0 — Cold
10012727 (Gastrointestinal disorders) | 0 | 2 | 0 | 0 — Diarrhea
10013036 (Eye disorders) | 1 | 0 | 0 | 0 — Diplopia
10013573 (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 — Dizziness
10013582 (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 — Dizziness
10013774 (Eye disorders) | 1 | 0 | 0 | 0 — Dry eye
10013786 (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — Dry skin
10013877 (Vascular disorders) | 0 | 1 | 0 | 0 — Deep vein thrombosis
10014542 (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — Emesis
10015573 (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — Acne
10015988 (Eye disorders) | 0 | 1 | 0 | 0 — Eyelid infection
10016791 (Infections and infestations) | 1 | 0 | 0 | 0 — Influenza like illness
10016952 (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Food poisoning
10017853 (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — Gastritis
10019044 (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — Hair Growth on face
10019045 (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — Hair loss
10019211 (Nervous system disorders) | 1 | 0 | 1 | 0 — Headache
10019428 (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 — Hematoma
10019523 (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — Hemoptysis
10021018 (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 — hypokalemia
10021143 (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — Hypoxia
10021282 (Nervous system disorders) | 1 | 0 | 0 | 0 — IIIrd nerve paralysis
10021680 (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Dyspnoea
10022437 (Psychiatric disorders) | 0 | 1 | 0 | 0 — Insomnia
10023086 (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 — Pruritus
10023090 (Eye disorders) | 0 | 1 | 0 | 0 — Eye pruritus
10023222 (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — joint pain
10027192 (Nervous system disorders) | 1 | 0 | 0 | 0 — Meningioma benign
10028050 (General disorders) | 0 | 2 | 0 | 0 — Abnormal MRI
10029410 (General disorders) | 2 | 2 | 0 | 0 — Night sweats
10033411 (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 — Arthralgia
10033432 (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 — Pain in hip
10033557 (Cardiac disorders) | 0 | 1 | 1 | 0 — Palpitations
10033733 (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — Papule (on chin)
10034474 (Cardiac disorders) | 0 | 1 | 0 | 0 — Pericardial Effusion
10036653 (General disorders) | 1 | 0 | 0 | 0 — Presyncope
10037402 (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — PH worsening
10037844 (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — Rash
10039792 (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 — Seborrhoea (oily hair)
10040604 (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — Shortness of breath
10042702 (General disorders) | 0 | 0 | 0 | 1 — Peripheral swelling
10046300 (Infections and infestations) | 0 | 1 | 0 | 0 — Upper respiratory tract infection
10046901 (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 — Vaginal discharge
10047115 (Vascular disorders) | 0 | 1 | 0 | 0 — Vasculitis
10049201 (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — Rash
10049498 (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — Pulmonary mass
10051626 (Eye disorders) | 1 | 0 | 0 | 0 — Conjunctivitis bacterial
10051792 (Product Issues) | 1 | 0 | 0 | 0 — Device Failure
10056739 (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — WBC increased
10059294 (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 — Seborrhoea
10059295 (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — Dry/Itchy Scalp
10073974 (Product Issues) | 0 | 1 | 0 | 0 — Device dislocation
10077730 (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Clinical Worsening - Change in WHO functional class
10080818 (General disorders) | 0 | 1 | 0 | 0 — Peripheral swelling

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT03648385/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT03648385/ICF_002.pdf